CLINICAL TRIAL: NCT04226625
Title: A Comparison of the Anesthetic and Hemodynamic Effects of a Volatile Anesthetic (Desflurane) and an Intravenous Anesthetic (Propofol), During Lung Volume Reduction Surgery
Brief Title: Effects of Desflurane and Propofol During Lung Volume Reduction Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAR3687; 9340 (Other: CPMC IRB)
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Lung Volume Reduction Surgery
Keywords: Anesthesia
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Intervention Model Description: Patients were randomized to receive propofol or desflurane as the maintenance anesthetic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Active Comparator): Patients will receive Propofol as an intravenous (IV) agent, which is administered into a vein through an IV line as a continuous infusion.
  Interventions: Drug: Propofol
- Desflurane (Active Comparator): Patients will receive Desflurane as a gas that is administered through an anesthesia machine.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — Intravenous administration
  Other Names: Diprivan
  Arms: Propofol
Drug: Desflurane — Volatile administration
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
Patients presenting for lung volume reduction are very high risk patients and it is important they receive the best anesthetic available. This study aims to answer which is the best anesthetic for managing such cases.

DETAILED DESCRIPTION:
The anesthetic technique for lung volume reduction surgery consists of a thoracic epidural in combination with a general anesthetic. The thoracic epidural is routine for this operation and allows administration of local anesthetics and painkillers in the epidural space which results in profound pain relief in the area of surgery. The epidural is routinely used for pain control during the surgery and after the surgery when the patient is awake.

The general anesthetic used may be a volatile agent (gas for example Desflurane), which is administered through the anesthesia machine, or an intravenous anesthetic agent, which is administered into a vein through an intravenous line as a continuous infusion (example Propofol). The use of an anesthetic agent and an epidural often causes a decrease in blood pressure which is treated with medication. The investigators are comparing the two anesthetic techniques regarding their effect on blood pressure and the amount of medication needed to treat it.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo lung volume reduction surgery (LVRS)

Exclusion Criteria:

* Does not sign a study consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-01-31 (Actual); Primary Completion 2001-03-21 (Actual); Study Completion 2002-03-21 (Actual)

PRIMARY OUTCOMES:
Time of discontinuation of anesthetic to eye opening | Up to 30 minutes (during procedure)
  Measured in minutes
Time of discontinuation of anesthetic to tidal volume (TV) 300ml | Up to 30 minutes (during procedure)
  Measured in minutes
Time of discontinuation of anesthetic to extubation | Up to 30 minutes (during procedure)
  Measured in minutes

SECONDARY OUTCOMES:
Duration of intensive care unit (ICU) stay | Up to 1 month from procedure
  Measured in days
Duration of hospital stay | Up to 1 month from procedure
  Measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Bessie Kachulis, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No